CLINICAL TRIAL: NCT04486209
Title: Non-invasive Spinal Cord Stimulation for Spasticity Control and Augmentation of Voluntary Motor Control in Individuals With Multiple Sclerosis
Acronym: noSpasMS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Neurological Center, Otto Wagner Hospital (Unknown)
Responsible Party: Principal Investigator, Ursula Hofstoetter, Senior researcher, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Version MS_tSCS_v1
Record Dates: First submitted 2020-07-17; First posted 2020-07-24 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Multiple Sclerosis
Keywords: neuromodulation; spinal cord stimulation; walking function; spasticity
MeSH Terms: conditions — Multiple Sclerosis; Muscle Spasticity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: transcutaneous spinal cord stimulation — electrical stimulation of the lumbosacral spinal cord through surface electrodes

SUMMARY:
Epidural spinal cord stimulation (SCS) is currently regarded as one of the most promising intervention methods to improve motor function in individuals with severe spinal cord injury. In parallel, an increasing number of studies is suggesting that noninvasive SCS can improve spasticity and residual motor control in the same subject population. The present study explores whether single sessions of noninvasive SCS would improve walking performance and ameliorate spasticity in individuals with multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of relapsing-remitting, primary- or secondary-progressive MS
* lower-limb spasticity

Exclusion Criteria:

* acute relapse of MS
* other neuromuscular diseases
* active and passive implants at vertebral level T9 or caudally
* dermatological issues at stimulation site
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-12-27 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2020-07-02 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth Scale | 24 hours

SECONDARY OUTCOMES:
10-m walk test | 24 hours
2-min walk test | 24 hours
Timed up an go test | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No